CLINICAL TRIAL: NCT01677897
Title: Impact of the Addition of Metformin to Abiraterone in Pre-docetaxel Metastatic Castration-resistant Prostate Cancer Patients Progressing on Abiraterone Treatment (MetAb-Pro): a Phase II Pilot Study
Brief Title: Impact of the Addition of Metformin to Abiraterone in Metastatic Prostate Cancer Patients
Acronym: MetAb-Pro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kantonsspital Graubünden (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Principal Investigator, Michael Mark, assistant medical director, Kantonsspital Graubünden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MetAb-Pro
Record Dates: First submitted 2012-08-28; First posted 2012-09-03 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin; abiraterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Metformin 2x1000mg orally per day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Adding Metformin to Abiraterone in case of PSA-Progression
  Other Names: Abiraterone

SUMMARY:
The purpose of this study is to assess the impact of the addition of metformin to abiraterone on survival in patients with metastatic prostate cancer

DETAILED DESCRIPTION:
The purpose of this study is to assess the impact of the addition of metformin to abiraterone on survival in patients with metastatic chemotherapy-naive prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Metastatic adenocarcinoma of the prostate.
* Patient must give written informed consent before registration.
* Age ≥18 years.
* WHO performance status 0-2.
* Tumor progression (as defined below) after at least 1 hormonal treatment (orchiectomy, LHRH agonist) with documented total testosterone levels ≤ 1.7 nmol/L (≤ 50 ng/dL). Ongoing concurrent use of LHRH agonist is required if the patient has not been surgically castrated.
* PSA progression during treatment with abiraterone (at least 12 weeks of treatment) defined as follows:

  * In case PSA levels had not decreased under treatment: ≥ 25% increase over baseline (at registration) AND an increase in the absolute PSA value of ≥ 5 ng/mL.
  * In case of PSA response < 50% under treatment: ≥ 25% increase over the nadir AND an increase in the absolute PSA value of ≥ 5 ng/mL.
  * In case of PSA response ≥ 50% under treatment: ≥ 50% increase over the nadir AND an increase in the absolute PSA value of ≥ 5 ng/mL Note: PSA progression has to be confirmed at least 1 week later. In case of confirmation the first date of PSA rise is relevant for the calculation.
* Serum potassium ≥ 3.5mmol/L.
* Adequate hematological values: neutrophils ≥1.5x109/L, platelets ≥100x109/L.
* Adequate hepatic function: bilirubin ≤1.5 x ULN, ALT ≤2.5 x ULN.
* Adequate renal function (calculated creatinine clearance ≥50 mL/min, according to the formula of Cockcroft-Gault).
* Able to swallow study drug as whole tablet.
* Patient compliance and geographic proximity allow proper staging and follow-up.

Exclusion Criteria:

* Previous malignancy within 2 years with the exception of localized non-melanoma skin cancer and Ta and Tis bladder cancer.
* Known CNS or spinal cord metastases.
* Active autoimmune disease requiring higher doses of corticosteroid than the equivalent of prednisone 10mg/d.
* Radiotherapy within the last 2 weeks before start of the trial treatment.
* Patients treated with anti-androgens such as flutamide or bicalutamide, if not discontinued at least 4 weeks prior to registration in case of response or in case of no response 2 weeks prior to inclusion for wash-out reasons.
* Prior treatment with metformin Prior treatment with metformin
* Diabetic ketoacidosis, diabetic coma and precoma
* Concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days prior to trial entry, except treatment with bisphosphonates and LHRH agonists.
* Known hypersensitivity to trial drugs or hypersensitivity to any of their components.
* Concomitant drugs contraindicated for use with the trial drugs according to the Swissmedic-approved product information.
* Uncontrolled hypertension, history of cardiac failure NYHA class III or IV.
* Serious underlying medical condition (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial (e.g. uncontrolled or acute severe infection, uncontrolled diabetes).
* Active or symptomatic viral hepatitis or chronic liver disease.
* History of pituitary or adrenal dysfunction.
* Gastrointestinal disorder affecting absorption.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, or interfering with compliance for oral drug intake.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
progression free survival | at 12 weeks

SECONDARY OUTCOMES:
overall survival | up to 2 years

OTHER OUTCOMES:
progression free survival at 24 weeks | at 24 weeks
progression free survival | up to 24 weeks
psa response | at 12 weeks
number of adverse events according to the NCI CTCAE v4.0 | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: michael mark, md, Principal Investigator — Kantonsspital Graubünden
Locations (1):
- Kantonsspital Graubünden, Chur, Kanton Graubünden, Switzerland

REFERENCES:
- [Derived] Mark M, Klingbiel D, Mey U, Winterhalder R, Rothermundt C, Gillessen S, von Moos R, Pollak M, Manetsch G, Strebel R, Cathomas R. Impact of Addition of Metformin to Abiraterone in Metastatic Castration-Resistant Prostate Cancer Patients With Disease Progressing While Receiving Abiraterone Treatment (MetAb-Pro): Phase 2 Pilot Study. Clin Genitourin Cancer. 2019 Apr;17(2):e323-e328. doi: 10.1016/j.clgc.2018.12.009. Epub 2019 Jan 2. PMID 30686756